CLINICAL TRIAL: NCT05091619
Title: A Randomized, Blinded, Parallel Controlled Phase 3 Clinical Study to Evaluate the Safety and Immunogenicity of the Diphtheria, Tetanus and Three-components Acellular Pertussis Combined Vaccine, Adsorbed in Healthy Infants at the Age of 2 Months and 3 Months
Brief Title: A Phase 3 Study of BIBP Diphtheria, Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed
Acronym: DTaP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Beijing Institute of Biological Products Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016L10765-2
Record Dates: First submitted 2021-10-21; First posted 2021-10-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-11

CONDITIONS: Whooping Cough; Diphtheria; Tetanus
MeSH Terms: conditions — Whooping Cough; Diphtheria; Tetanus | interventions — Tetanus Toxoid; Vaccines, Combined; Pentavac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- A1 (Experimental): subjects aged 3 months receive 3 doses of vaccines with a interval of 30 days for primary immunization, and a booster dose at 18 month old
  Interventions: Biological: Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed
- A2 (Active Comparator): subjects aged 3 months receive 3 doses of vaccines with a interval of 30 days for primary immunization, and a booster dose at 18 month old
  Interventions: Biological: Diphtheria,Tetanus and Acellular Pertussis Combined Vaccine, Adsorbed
- A3 (Active Comparator): subjects aged 3 months receive 3 doses of vaccines with a interval of 30 days for primary immunization, and a booster dose at 18 month old
  Interventions: Biological: Diphtheria,tetanus,pertussis(acellular,component),poliomyelitis(inactivated) vaccine(absorbed) and Haemophilus influenzae type b conjugate vaccine
- B1 (Experimental): subjects aged 2 months receive 3 doses of vaccines with a interval of 30 days for primary immunization, and a booster dose at 18 month old
  Interventions: Biological: Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed
- B2 (Active Comparator): subjects aged 2 months receive 3 doses of vaccines with a interval of 30 days for primary immunization, and a booster dose at 18 month old
  Interventions: Biological: Diphtheria,Tetanus and Acellular Pertussis Combined Vaccine, Adsorbed
- B3 (Experimental): subjects aged 2 months receive 3 doses of vaccines with a interval of 2 months for primary immunization, and a booster dose at 18 month old
  Interventions: Biological: Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed
- C1 (Experimental): subjects aged 3 months receive 3 doses of lot-1 vaccines with a interval of 30 days for primary immunization
  Interventions: Biological: Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed
- C2 (Experimental): subjects aged 3 months receive 3 doses of lot-2 vaccines with a interval of 30 days for primary immunization
  Interventions: Biological: Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed
- C3 (Experimental): subjects aged 3 months receive 3 doses of lot-3 vaccines with a interval of 30 days for primary immunization
  Interventions: Biological: Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed

INTERVENTIONS:
Biological: Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed — Intramuscular injection
  Other Names: DTacP
  Arms: A1; B1; B3; C1; C2; C3
Biological: Diphtheria,Tetanus and Acellular Pertussis Combined Vaccine, Adsorbed — Intramuscular injection
  Other Names: DTaP
  Arms: A2; B2
Biological: Diphtheria,tetanus,pertussis(acellular,component),poliomyelitis(inactivated) vaccine(absorbed) and Haemophilus influenzae type b conjugate vaccine — Intramuscular injection
  Other Names: PENTAXIM
  Arms: A3

SUMMARY:
The study will evaluate the safety, immunogenicity，immune persistence and lot-to-lot consistency of Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed, (DTacP) including 2 parts:

PART 1 will evaluate the safety and immunogenicity of DTacP in health infants aged 2 months and 3 months compared with an adsorption Tetanus-diphtheria-acellular Pertussis (DTaP) Vaccine and Diphtheria,tetanus,pertussis(acellular,component),poliomyelitis(inactivated) vaccine(absorbed) and Haemophilus influenzae type b conjugate vaccine (PENTAXIM)，compare the safety and immunogenicity of DTacP with different immunization schedules, and observe the immune persistence.

PART 2 will evaluate the lot-to-lot consistency of DTacP in health infants aged 3 months with the 3-dose schedule of 3-4-5 month.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 2months (60-89 days) and 3months (90-119 days) ；
* Willing to provide proof of identity
* Subjects aged 2 months have not been vaccinated with DTaP, IPV, Hib, or 13-valent pneumococcal polysaccharide conjugate vaccine;
* Subjects of 3 months have not been inoculated with DTaP vaccine, and IPV (only group A3）；
* Subjects'guardians or trustees are able to understand and sign the informed consent voluntarily, comply with the requirements of the clinical study plan.

Exclusion Criteria:

* With temperature >37.0°C on axillary setting before vacciation;
* With a medical history of diphtheria, pertussis or tetanus;
* Had contact with individuals with confirmed pertussis, diphtheria and tetanus diseases in their families in the past 30 days;
* Premature birth (delivery before the 37th week of pregnancy)or low birth weight (birth weight< <2500g);
* History of dystocia, suffocation rescue, neurological damage;
* With congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* History of epilepsy, convulsions or convulsions, or have a family history of mental illness;
* History of abnormal blood coagulation (such as coagulation factor deficiency, coagulopathy);
* Had received immune enhancement or inhibitor therapy (continuous oral or instillation for more than 14 days);
* History of severe allergic reactions to vaccination, such as difficulty breathing, urticaria;
* Any prior administration of blood products in last 3 month;
* Any prior administration of attenuated live vaccine in last 14 days;
* Any prior administration of subunit or inactivated vaccines in last 7 days;
* Plans to participate in or is participating in any other drug clinical study;
* Has any other factors judged by investigators that make them unfit to participate in the clinical trial

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2898 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2027-09-22 (Estimated)

PRIMARY OUTCOMES:
The seroconversion rate of anti-pertussis toxoid , anti-filamentous hemagglutinin, anti-Pertactin, anti-diphtheria toxoid and anti-tetanic antibody | 1 month after Dose 3
  seroconversion is defined as post-third dose antibody concentrations ≥ protective antibody concentration if pre-vaccination concentration is < protective antibody concentration, or ≥ 4 x protective antibody concentration if pre-vaccination concentrations ≥ protective antibody concentration.
Geometric Mean Concentrations (GMCs) of anti-pertussis toxoid , anti-filamentous hemagglutinin, anti-Pertactin, anti-diphtheria toxoid and anti-tetanic antibody | 1 month after Dose 3
  As measured at the central laboratory
Percentage of participants reporting local reactions | Day 7 post-each dose
  As elicited by investigational site staff
Percentage of participants reporting systemic events | Day 7 post-each dose
  As elicited by investigational site staff
Percentage of participants reporting adverse events | within 30 days post-each dose
  As elicited by investigational site staff

SECONDARY OUTCOMES:
The seropositivity rate of anti-pertussis toxoid , anti-filamentous hemagglutinin, anti-Pertactin, anti-diphtheria toxoid and anti-tetanic antibody | Day 30 post-dose 3
  Seropositivity is defined as post-3 dose antibody concentrations ≥ protective antibody concentration
Geometric Mean Concentrations (GMCs) of anti-pertussis toxoid , anti-filamentous hemagglutinin, anti-Pertactin, anti-diphtheria toxoid and anti-tetanic antibody | before dose 4 at 18 months old(booster)
  As measured at the central laboratory
The seropositivity rate of anti-pertussis toxoid , anti-filamentous hemagglutinin, anti-Pertactin, anti-diphtheria toxoid and anti-tetanic antibody | before dose 4 at 18 months old(booster)
  Seropositivity is defined as antibody concentrations ≥ protective antibody concentration
Geometric Mean Concentrations (GMCs) of anti-pertussis toxoid , anti-filamentous hemagglutinin, anti-Pertactin, anti-diphtheria toxoid and anti-tetanic antibody | Day 30 post-dose 4 at 18 months old(booster)
  As measured at the central laboratory
The seropositivity rate of anti-pertussis toxoid , anti-filamentous hemagglutinin, anti-Pertactin, anti-diphtheria toxoid and anti-tetanic antibody | Day 30 post-dose 4 at 18 months old(booster)
  eropositivity is defined as antibody concentrations ≥ protective antibody concentration

OTHER OUTCOMES:
Geometric Mean Concentrations (GMCs) of anti-pertussis toxoid , anti-filamentous hemagglutinin, anti-Pertactin, anti-diphtheria toxoid and anti-tetanic antibody | 12th month, 24th month, 36th month post-dose 4 , before 6 years old and day 30 post-dose 5
  As measured at the central laboratory
The seropositivity rate of anti-pertussis toxoid , anti-filamentous hemagglutinin, anti-Pertactin, anti-diphtheria toxoid and anti-tetanic antibody | 12th month, 24th month, 36th month post-dose 4 , before 6 years old and day 30 post-dose 5
  Seropositivity is defined as antibody concentrations ≥ protective antibody concentration

CONTACTS AND LOCATIONS:
Overall Officials: Lili Huang, Principal Investigator — Henan Province Center for Disease Control and Prevention
Locations (4):
- China (4):
  - Neihuang County Center for Disease Control and Prevention, Anyang, Henan
  - Wen County Center for Disease Control and Prevention, Jiaozuo, Henan
  - Wuyang County Center for Disease Control and Prevention, Luohe, Henan
  - Yanjin County Center for Disease Control and Prevention, Xinxiang, Henan

IPD SHARING:
Plan to Share IPD: No
In order to maintain the rights of the subject, do not open the IPD